CLINICAL TRIAL: NCT07050927
Title: Long-Term Effect of Online Occupational Therapy-Based Parent Training on Feeding Problems in Infants: A Randomized Controlled Longitudinal Study
Brief Title: Long-Term Effect of Online Occupational Therapy-Based Parent Training on Feeding Problems in Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Rukiye Begüm KOCA, Lecturer Rukiye Begüm Koca Şentürk, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Decision No: 112
Record Dates: First submitted 2025-06-22; First posted 2025-07-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Feeding Difficulties; Feeding Problems; Food Neophobia
Keywords: pediatrics; early childhood; telerehabilitation; parent training; group training; occupational therapy; feeding; feeding difficulties; feeding problems
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Training Group (Experimental): Participants in this group will receive a 4-week online occupational therapy-based parent training via secure Zoom sessions. The training focuses on feeding skills development, sensory strategies, parenting attitudes, and stress management. Participants will complete assessments at baseline, 6 months, and 12 months using standardized tools to evaluate infant feeding behavior, parental attitudes, and parenting stress
  Interventions: Behavioral: Online occupational therapy group training
- Non-intervention Group (No Intervention): Participants in this group will not receive any intervention during the study period. They will complete the same assessments as the intervention group at baseline, 6 months, and 12 months to monitor changes in infant feeding behavior, parental attitudes, and parenting stress.

INTERVENTIONS:
Behavioral: Online occupational therapy group training — The intervention is a 4-week online parent training program based on occupational therapy principles, delivered via secure Zoom sessions once per week. Each session lasts approximately 60-75 minutes and focuses on topics such as feeding skill development, sensory-based feeding difficulties, responsive parenting strategies, and stress management techniques. The training includes interactive discussions and practical suggestions for daily feeding routines. Supporting materials, such as PDF slides and short demonstration videos, are shared with participants after each session. Attendance in at least three sessions is required to remain in the study.
  Arms: Parent Training Group

SUMMARY:
This study type is a clinical trial (randomized controlled longitudinal study). The primary purpose is to determine whether an online occupational therapy-based parent training program can prevent or reduce feeding problems, improve parental attitudes, and decrease parenting stress in mothers of infants.

The participant population includes female caregivers (mothers) of typically developing infants aged 18 to 24 months. All participants are healthy volunteers.

The main research questions this study aims to answer are:

Does online occupational therapy-based parent training reduce feeding problems in infants (e.g., food refusal, resistance, sensory-based rejection)? Does the training improve maternal attitudes related to feeding and reduce parenting-related stress? Comparison group: Researchers will compare the outcomes of mothers who receive the online training (intervention group) with those who receive no intervention (control group) to determine the effectiveness of the program.

Participants will be asked to:

Complete baseline assessment forms prior to randomization

If in the intervention group:

Attend a 4-week online group training program (one session per week) via a secure Zoom® platform Participate in follow-up assessments at 6 months and 12 months post-training

All participants (in both groups) will:

Complete standardized assessment tools at three time points (baseline, 6-month follow-up, 12-month follow-up), including:

Sociodemographic Information Form Infant Adaptive Feeding Behavior Scale Feeding Process Parental Attitude Scale Parenting Stress Scale

ELIGIBILITY:
Inclusion Criteria:

* Mothers of typically developing infants aged between 18 and 24 months
* Mothers who report a stress level of 7 or above on a visual analog scale regarding their child's feeding process
* Mothers who have the necessary technical equipment to follow the occupational therapy training via online platforms

Exclusion Criteria:

* Infants born prematurely or diagnosed with significant neurological or developmental conditions
* Infants who receive any diagnosis during the intervention or follow-up period
* Mothers in the intervention group who miss more than one training session
* Mothers who are currently receiving or have previously received occupational therapy or feeding counseling

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Individuals who identify as the mother or primary female caregiver of a typically developing infant aged 18-24 months are eligible to participate.
Enrollment: 32 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Adaptive Eating Behavior in Infancy Scale | T₀ - Baseline: Pre-training, first assessment after randomization T₁ - Post-intervention: Immediately after training completion T₂ - 6-month follow-up T₃ - 12-month follow-up
  The Infant Adaptive Feeding Behavior Scale (IAFBS) was developed by Dilsiz and Dağ in 2018 to assess the eating behaviors of children aged 9 to 36 months. The scale consists of 20 items and four factors: "Reluctance," "Resistance," "Reaction to Main Meal Structure," and "Sensory-Related Food Refusal." Items 1-8 measure the reluctance factor; items 9-12 measure resistance; items 13-16 assess reactions to meal structure; and items 17-20 evaluate food refusal related to sensory issues.
  Items are rated on a 5-point Likert scale ranging from "Never" to "Always," scored as follows: never = 1, rarely = 2, sometimes = 3, usually = 4, always = 5. However, item 2 ("reaches spontaneously for food during meals") reflects a positive feeding behavior and is reverse-scored. All other items are scored in the standard direction.
  The total score ranges from 20 to 100. Higher total and subscale scores indicate more severe feeding behavior problems in infants aged 9 to 36 months.
Maternal Attitudes Scale in the Feeding Process | T₀ - Baseline: Pre-training, first assessment after randomization T₁ - Post-intervention: Immediately after training completion T₂ - 6-month follow-up T₃ - 12-month follow-up
  This scale was developed in 2018 by Dilsiz and Dağ with the aim of identifying problematic areas in maternal attitudes during the feeding process, based on the interactional dimension of feeding between the mother and child. The Feeding Process Parental Attitude Scale (FPPAS) is used to assess the feeding-related attitudes of mothers with children aged 9 to 72 months. It is a 5-point Likert-type scale with response options ranging from "Never" to "Always." The scale consists of 27 items and includes the following subscales: Negative Emotional State During Meals, Attitudes Toward Inadequate/Unbalanced Nutrition, Negative Feeding Strategies, Forceful Feeding, and Reaction to Others' Opinions. The total score ranges from 27 to 135. Higher scores on the total scale and subscales indicate a greater presence of problematic maternal attitudes regarding the feeding process.
Parental Stress Scale | T₀ - Baseline: Pre-training, first assessment after randomization T₁ - Post-intervention: Immediately after training completion T₂ - 6-month follow-up T₃ - 12-month follow-up
  The Parenting Stress Scale was developed by Aydoğan and Özbay in 2017 to measure the stress experienced by parents of typically developing children in relation to their parenting role. The scale consists of 18 items and has a single-factor structure that includes the parent, the parent-child relationship, and characteristics of the child. It is a Likert-type instrument rated from 0 ("Does not describe at all") to 4 ("Describes very well"). The total score ranges from 0 to 72, with higher scores indicating higher levels of parenting stress. The scale is easily applicable to parents who have at least one child and have completed primary education or higher.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect participant confidentiality and comply with ethical standards.